CLINICAL TRIAL: NCT00246636
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase IV Study to Assess the Efficacy and Safety of Adjunctive Omacor Therapy in Hypertriglyceridemic Subjects Treated With Antara, Followed by an 8-week Extension
Brief Title: Evaluation of Efficacy and Safety of Omacor (Omega-3-acid Ethyl Esters) as Add-on Therapy in Hypertriglyceridemic Subjects Treated With Antara (Fenofibrate) Followed by an 8-week Extension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OM5 program (Reliant); OM5/LOV111859 (original study); OM5X/LOV111860 (1st extension)
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Last update posted 2009-12-14 (Estimated); Status verified 2009-12

CONDITIONS: Hypertriglyceridemia
Keywords: Very high triglycerides; omega-3-acid ethyl esters; fenofibrate; Lovaza
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Fenofibrate; Omacor

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- OM5/LOV111859 (double-blind study) - Antara (Active Comparator): Antara (fenofibrate) + placebo
  Interventions: Drug: Antara (fenofibrate)
- OM5X/LOV111860 (extension study) - Open-Label Antara + Lovaza (Experimental): Open-label Antara (fenofibrate) + Lovaza (omega-3-acid ethyl esters) [formerly known as Omacor]
  Interventions: Drug: Antara (fenofibrate) + Lovaza; Drug: Antara (fenofibrate)
- OM5/LOV111859 (double-blind study) - Antara + Lovaza (Experimental): Antara (fenofibrate) + Lovaza (omega-3-acid ethyl esters) [formerly known as Omacor]
  Interventions: Drug: Antara (fenofibrate) + Lovaza

INTERVENTIONS:
Drug: Antara (fenofibrate) + Lovaza — Antara (fenofibrate) + Lovaza (omega-3-acid ethyl esters) [formerly known as Omacor]
  Arms: OM5/LOV111859 (double-blind study) - Antara + Lovaza; OM5X/LOV111860 (extension study) - Open-Label Antara + Lovaza
Drug: Antara (fenofibrate) — Antara (fenofibrate) + placebo
  Arms: OM5/LOV111859 (double-blind study) - Antara; OM5X/LOV111860 (extension study) - Open-Label Antara + Lovaza

SUMMARY:
The purpose of OM5/LOV111859 was to evaluate efficacy and safety of Omacor (omega-3-acid ethyl esters) as add-on therapy to Antara (fenofibrate) and diet for the treatment of patients with very high triglycerides.

The purpose of both OM5X/LOV111860 was to assess the continued efficacy and safety of adjunctive Lovaza (omega-3-acid ethyl esters) therapy in hypertriglyceridemic subjects treated with fenofibrate in lowering serum triglyceride (TG) levels.

DETAILED DESCRIPTION:
Three studies comprise this OM5 Program

* Study OM5 / LOV111859 (double-blind study) and OM5X / LOV111860 (1st open-label extension) are part of this listing on ClinicalTrials.gov - NCT00246636.
* Study OM5XX / LOV111821 (2nd open-label extension) is listed as a separate listing on ClinicalTrials.gov - NCT00891293

ELIGIBILITY:
For OM5/LOV111858 -

Inclusion Criteria:

* Men and women ages 18-79 years, inclusive
* Triglyceride levels between 500 mg/dL and <1300 mg/dL
* Body mass index between 25 and 43 kg/m2
* Willingness to follow a low-saturated fat diet during the study period and maintain current physical activity level
* Normally active and in good health on the basis of medical history, brief physical examination, electrocardiogram, and routine laboratory tests
* Provide written informed consent and authorization for protected health information disclosure

Exclusion Criteria:

* Sensitivity to fibrate drugs or omega-3 fatty acids
* Lipoprotein lipase impairment or apo C-2 deficiency or Type III hyperlipidemia
* History of pancreatitis
* Recent history of certain kidney, liver, lung, or gastrointestinal disease or cancer (except non-melanoma skin cancer)
* Poorly controlled diabetes mellitus
* Type 1 diabetes
* Pregnant or lactating females. Women of childbearing potential who are not using a medically approved method of contraception.
* Use of certain types of hormones, anticonvulsant drugs, immunologic drugs, antibiotic, antifungal and antiviral drugs, and cardiac drugs
* Use of isotretinoin (Accutane)
* Use of warfarin (Coumadin)

For OM5X/LOV111859 -

Subjects were included in the study if they met the following criteria:

1. Satisfied all inclusion and exclusion criteria prior to and throughout the previous OM5 study or had a corresponding approved protocol deviation
2. Successfully completed the previous OM5 double-blind study to Week 8
3. Provided written informed consent on or before the Week 8 clinic visit of the OM5 double-blind study (i.e., Visit 1X of the OM5X extension study)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2005-10; Primary Completion 2007-02 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
OM5X/LOV111860 - Difference between double-blind Lovaza (omega-3-acid ethyl esters) + fenofibrate (Group 1) and placebo + fenofibrate (Group 2) treatment groups in percent change in fasting serum TG level from baseline of OM5 to end of OM5X | 8 weeks
OM5/LOV111859 - Difference between Lovaza (omega-3-acid ethyl esters) [formerly known as Omacor]+ fenofibrate and placebo + fenofibrate treatment groups in percent change in TG level from baseline | 8 weeks

SECONDARY OUTCOMES:
OM5X/LOV111860 - Difference between double-blind Lovaza (omega-3-acid ethyl esters) + fenofibrate (Group 1) and placebo + fenofibrate (Group 2) treatment groups in percent change for other lipid and biomarkers from baseline of OM5 to end of OM5X | 8 weeks
OM5/LOV111859 - Difference between Lovaza (omega-3-acid ethyl esters) + fenofibrate and placebo + fenofibrate treatment groups in percent change for other lipid and biomarkers from baseline | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Bays HE, Maki KC, Doyle RT, Stein E. The effect of prescription omega-3 fatty acids on body weight after 8 to 16 weeks of treatment for very high triglyceride levels. Postgrad Med. 2009 Sep;121(5):145-50. doi: 10.3810/pgm.2009.09.2061. PMID 19820283
- [Derived] Roth EM, Bays HE, Forker AD, Maki KC, Carter R, Doyle RT, Stein EA. Prescription omega-3 fatty acid as an adjunct to fenofibrate therapy in hypertriglyceridemic subjects. J Cardiovasc Pharmacol. 2009 Sep;54(3):196-203. doi: 10.1097/FJC.0b013e3181b0cf71. PMID 19597368